CLINICAL TRIAL: NCT00682890
Title: Combination Metformin and Oral Contraception for Polycystic Ovary Syndrome (PCOS)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R03HD047298 (NIH)
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Polycystic Ovary Syndrome; PCOS; Insulin Sensitivity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo tablet and birth control pill daily
  Interventions: Drug: placebo
- 2 (Active Comparator): metformin 2000 mg and birth control pill daily
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: placebo — placebo birth control pill daily
  Arms: 1
Drug: metformin — 2000 mg per day for 3 months daily birth control pill
  Arms: 2

SUMMARY:
The purpose of this research study is to determine if adding Metformin, a drug that reduces insulin resistance, to birth control pills will reduce the risk of developing type 2 diabetes, high blood pressure. high lipid levels and heart disease in women with PCOS

DETAILED DESCRIPTION:
Inclusion criteria: PCOS women between the ages of 18-45,< 8 periods annually, elevated serum free testosterone, normal thyroid function tests and serum prolactin, exclusion of late onset adrenal hyperplasia, acceptable health based on interview and medical history, physical exam and lab tests, ability to comply with the requirements of the study and to provide signed, witnessed informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-45, , 8 menstrual cycles annually, elevated serum free testosterone, normal thyroid function test and serum prolactin, exclusion of late onset adrenal hyperplasia

Exclusion Criteria:

* Diabetes mellitus, pulmonary, cardiac, renal, hepatic, cholestatic, neurologic, psychiatric, infectious, malignant diseases,history of breast cancer, history of Deep Vein Thrombosis, pregnancy and lactation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2005-11; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Dunn, MD, Study Director — DSMB
Locations (1):
- General Clinical Research Center, Richmond, Virginia, United States

REFERENCES:
- [Result] Essah PA, Arrowood JA, Cheang KI, Adawadkar SS, Stovall DW, Nestler JE. Effect of combined metformin and oral contraceptive therapy on metabolic factors and endothelial function in overweight and obese women with polycystic ovary syndrome. Fertil Steril. 2011 Aug;96(2):501-504.e2. doi: 10.1016/j.fertnstert.2011.05.091. Epub 2011 Jul 5. PMID 21733508
- See also: Related Info — http://www.vcu.edu/pcos

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment and testing conducted at VCU General Clinical Research Center from August 2006 to December 2009
Pre-assignment Details: Following enrollment but prior to group assignment 5 subject were excluded based on screening results. Randomized remaining 23 subjects.
Groups:
- Placebo: Placebo tablet and birth control pill daily
- Metformin: metformin 2000 mg and birth control pill daily
Period: Overall Study
Arm/Group | Placebo | Metformin
Started | 12 | 11
Completed | 10 | 9
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — subject moved away | 0 | 1
Not completed — heavy menstrual bleeding | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Metformin | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (1.3) | 26.6 (1.4) | 25.5 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 32.6 (2.3) | 36.2 (2.5) | 34.4 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity Measures: Insulin Sensitivity Index (ISI)
Description: Insulin sensitivity as measured by a combination of insulin sensitivity index (ISI) which should go up after 3 month treatment period to show improvement, and insulin sensitivity (SI) which should go down after 3 month treatment period to show improvement. Note that the ISI as developed by Matsuda and DeFronzo from a calculation based on results from a standard oral glucose tolerance test (OGTT) (doi: 10.2337/diacare.22.9.1462 Diabetes Care September 1999 vol. 22 no. 9 1462-1470) is recorded as units on an arbitrary scale. SI data is based on a calculation derived from analysis of results of frequently sampled intravenous glucose tolerance test (FSIVGTT) by Bergman et al (doi:10.1172/JCI112886/J Clin Invest. 1987;79(3):790-800) and is reported with units min-1/(µlU/L).
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 10 | 9
units on a scale
  ISI at baseline | 4.7 (1.6) | 7.3 (1.7)
  ISI at month 3 | 4.4 (0.96) | 5.9 (1.0)
  ISI change vs baseline | -0.3 (1.1) | -1.4 (1.2)
Statistical Analysis 1: Comparison: Placebo; P value on change at 3 months for placebo group; Test type: Superiority or Other; p = 0.63, ANOVA
Statistical Analysis 2: Comparison: Metformin; Test type: Superiority or Other; p = 0.42, ANOVA

2. Primary Outcome: Change in Insulin Sensitivity Measures: Insulin Sensitivity (SI)
Description: as for outcome 1
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: min-1/(µlU/L)
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 10 | 9
min-1/(µlU/L)
  SI at baseline | 2.26 (0.48) | 3.83 (0.78)
  SI at 3 months | 2.8 (0.87) | 2.11 (0.44)
  SI change vs baseline | 0.544 (0.79) | -1.72 (0.61)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p = 0.51, ANOVA
Statistical Analysis 2: Comparison: Metformin; Test type: Superiority or Other; p = 0.03, ANOVA

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Placebo | Metformin
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

LIMITATIONS AND CAVEATS:
study duration was relatively brief,earlier serum markers of the inflammatory process,e.g.,IL-6, were not evaluated,sample size planned was not achieved despite intensive recruitment efforts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No